CLINICAL TRIAL: NCT07133672
Title: The Effect of Digital Physiotherapy Practices on Pulmonary Functions, Respiratory Muscle Strength, Functional Capacity, Upper Extremity Peripheral Muscle Strength and Quality of Life in Patients Undergoing Thoracic Surgery
Brief Title: Effect of Digital Physiotherapy Practice on Pulmonary Function, Muscle Strength, Quality of Life After Thoracic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşegül Şahin, Physiotherapist, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BVUaysegul001
Record Dates: First submitted 2025-07-09; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Surgery
Keywords: Physiotherapy; Thoracic surgery; Exercises
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): During the initial face-to-face assessment session, patients will be provided with general information regarding key points to consider following thoracic surgery. Instruction on the proper techniques for performing breathing exercises will also be given. The exercise training sessions will be structured to include approximately 10 minutes of warm-up, around 30 minutes of goal-oriented exercises, and a final 10-minute cool-down period, resulting in a total average duration of 50 minutes per session.
  Interventions: Other: Exercise
- Control group (Active Comparator): During the initial face-to-face assessment session, patients will be provided with general information regarding key points to consider following thoracic surgery.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Exercise — Exercise sessions will begin with flexibility exercises targeting the shoulder and neck regions. This will be followed by breathing exercises utilizing fundamental respiratory techniques. Extremity exercises will include movements focused on the upper extremities and trunk, with progression applied according to a pre-established plan. Each session will conclude with cool-down exercises. Additionally, patients will be encouraged to engage in regular walking on a weekly basis.
  Arms: Training group
Other: Standard care — Patients will receive education regarding the critical aspects to consider after hospital discharge. Standard postoperative care protocols will be implemented.
  Arms: Control group

SUMMARY:
Thoracic surgery is the primary intervention used in the treatment of diseases affecting the lungs, pleura, chest wall, and mediastinum. Postoperative changes occur in both lung functions and clinical symptoms due to the procedure itself and patient-related factors. After thoracic surgery, patients often experience reduced exercise tolerance and impaired respiratory functions, negatively affecting their participation in daily activities, functional levels, and quality of life. In open thoracotomies, the incision site, severed muscles, and the size of the incision can impact upper extremity and trunk functions. The aim of this study is to investigate the effects of physiotherapy applied through digital methods on respiratory functions, respiratory muscle strength, functional capacity, upper extremity muscle strength, and quality of life in patients who have undergone thoracic surgery.

DETAILED DESCRIPTION:
Thoracic surgery is a primary intervention used in the treatment of diseases of the lungs, pleura, chest wall, and mediastinum. Following surgery, changes in lung function and associated clinical symptoms may occur due to both the surgical procedure itself and patient-specific factors, and these may present intraoperatively and/or postoperatively. These changes are primarily restrictive in nature and may include a characteristic reduction in lung volume, a decrease in functional residual capacity that may lead to atelectasis, slowed mucociliary clearance, gas exchange abnormalities, and especially reduced chest expansion on the operated side. Additionally, problems in surfactant production and diaphragmatic dysfunction may also arise. Furthermore, the use of surgical drains, the nature of the surgical procedure, the integrity of the remaining lung tissue after resection, and the limitations caused by enforced immobility can all contribute to the development of various postoperative complications. Preventing and/or managing these postoperative complications is essential for enabling the patient to return to functional life, reducing long-term healthcare utilization, and improving survival rates. For this reason, pulmonary rehabilitation is indicated after thoracic surgeries. One of the methods of delivering rehabilitation is telerehabilitation, which allows patients to access therapy remotely. In this study, however, the term Digital Physiotherapy, which is a more current and comprehensive term recommended by World Physiotherapy, will be used. In the literature review, it was observed that most postoperative studies following thoracic surgery focus on the in-hospital period, while studies conducted after discharge are usually of short duration. The aim of this study is to examine the effects of long-term physiotherapy delivered through digital methods following thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent open thoracotomy
* Agreement to participate in the study
* Being between the ages of 18-75
* Having an internet connection at home and being able to participate in video-conference sessions via desktop-laptop computers, smartphones, electronic tablets, etc.

Exclusion Criteria:

* Pneumonectomy surgeries
* Having a cardiac, orthopedic, neurological or systemic disease that would prevent exercise
* Having mental, communication or behavioral disorders that would cause problems in understanding commands and questions or performing exercises.
* Participating in a pulmonary rehabilitation program before surgery
* Having been hospitalized for any pulmonary disease during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 12 weeks
  The volume of air exhaled during a full and strongest exhalation possible after a full inspiration, as measured by a spirometry device.
Forced expiratory volume in 1 second (FEV1) | 12 weeks
  FEV1 is the expiratory volume in the first second of the FVC maneuver.
Tiffeneau ratio (FEV1/FVC) | 12 weeks
  The FEV1/FVC represents the fraction of air a patient exhales in the first second. This measurement is crucial for detecting airflow obstruction.
Peak expiratory flow (PEF) | 12 weeks
  Peak Expiratory Flow (PEF) is defined as a maximal expiratory flow generated during a simple maneuver using a peak flow meter via a mouthpiece.
Respiratory Muscle Strength | 12 weeks
  Maximum inspiratory and expiratory pressures are measured using an intraoral pressure measuring device.
Functional Capacity | 12 weeks
  Six-Minute Walking Test Distance measurement (in meter).
Upper Extremity Peripheral Muscle Strength | 12 weeks
  Measurement of shoulder flexion and abduction muscle strength using an electronic hand dynamometer.
Health Related Quality of Life | 12 weeks
  Saint George Respiratory Questionnaire Results. Scores range from 1 to 100. Higher scores mean worse health.

SECONDARY OUTCOMES:
Shoulder Joint Range of Motion Measurement | 12 weeks
  Change of shoulder flexion and abduction range of motion
Trunk Lateral Flexion Flexibility | 12 weeks
  It is the measurement of the distance between the first and last points during lateral flexion of the trunk with a tape measure. (in centimeters)
Chest Expansion | 12 weeks
  Evaluation of change in chest expansion. The largest differences between maximum inspiration and maximum expiration is recorded as chest expansion.
Shoulder Pain | 12 weeks
  Assessment is made using the Shoulder Pain and Disability Index. Higher scores indicate more severe pain and greater disability.
Sleep | 12 weeks
  Assessment is made using the Insomnia Severity Index. Scores range from 0-28. A score of 8 or above is considered insomnia.